CLINICAL TRIAL: NCT02918617
Title: Clinical Efficacy in Relieving Dentin Hypersensitivity of Nanohydroxyapatite-Containing Toothpastes and Cream
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Sangi Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Bennett Amaechi, Professor, Department of Comprehensive Dentistry, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC20150221H
Record Dates: First submitted 2016-09-13; First posted 2016-09-29 (Estimated); Results first posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Dentin Sensitivity
Keywords: dentin hypersensitivity; nanohydroxyapatite; calcium sodium phosphosilicate; toothpaste; tooth cream
MeSH Terms: conditions — Dentin Sensitivity | interventions — potassium nitrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (9):
- Control toothpaste containing Novamin® technology (Active Comparator): Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Interventions: Drug: Control toothpaste containing Novamin® technology
- Control toothpaste containing 1500 ppm fluoride as MFP (Placebo Comparator): Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Interventions: Drug: Control toothpaste containing 1500 ppm fluoride as MFP
- Test toothpaste with nano-HAP (high concentration) (Experimental): Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Interventions: Drug: Test toothpaste with nano-HAP (high concentration)
- Test toothpaste with nano-HAP (low concentration) (Experimental): Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Interventions: Drug: Test toothpaste with nano-HAP (low concentration)
- Test toothpaste with nano-HAP and potassium nitrate (KNO3) (Experimental): Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Interventions: Drug: Test toothpaste with nano-HAP and (Potassium Nitrate) KNO3
- Control toothpaste without nano-HAP (Placebo Comparator): Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Interventions: Drug: Control toothpaste without nano-HAP
- Test toothpaste with nano-HAP (medium concentration) (Experimental): Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Interventions: Drug: Test toothpaste with nano-HAP (medium concentration)
- Test cream with nano-HAP (higher concentration) (Experimental): Participants will be instructed to brush for 2 minutes morning and evening with a full ribbon of standard fluoride toothpaste. After the evening brushing, participants will then insert custom-made trays loaded with a full ribbon of cream. Participants will be instructed to remove the trays after 5 minutes and expectorate the cream. Participants will be instructed not to eat or drink until the next morning following cream use.
  Interventions: Drug: Test cream with nano-HAP (higher concentration)
- Control cream without nano-HAP (Placebo Comparator): Participants will be instructed to brush for 2 minutes morning and evening with a full ribbon of standard fluoride toothpaste. After the evening brushing, participants will then insert custom-made trays loaded with a full ribbon of cream. Participants will be instructed to remove the trays after 5 minutes and expectorate the cream. Participants will be instructed not to eat or drink until the next morning following cream use.
  Interventions: Drug: Control cream without nano-HAP

INTERVENTIONS:
Drug: Control toothpaste containing Novamin® technology
  Arms: Control toothpaste containing Novamin® technology
Drug: Control toothpaste containing 1500 ppm fluoride as MFP
  Arms: Control toothpaste containing 1500 ppm fluoride as MFP
Drug: Test toothpaste with nano-HAP (high concentration)
  Arms: Test toothpaste with nano-HAP (high concentration)
Drug: Test toothpaste with nano-HAP (low concentration)
  Arms: Test toothpaste with nano-HAP (low concentration)
Drug: Test toothpaste with nano-HAP and (Potassium Nitrate) KNO3
  Arms: Test toothpaste with nano-HAP and potassium nitrate (KNO3)
Drug: Control toothpaste without nano-HAP
  Arms: Control toothpaste without nano-HAP
Drug: Test toothpaste with nano-HAP (medium concentration)
  Arms: Test toothpaste with nano-HAP (medium concentration)
Drug: Test cream with nano-HAP (higher concentration)
  Arms: Test cream with nano-HAP (higher concentration)
Drug: Control cream without nano-HAP
  Arms: Control cream without nano-HAP

SUMMARY:
This study will investigate the effectiveness of nanohydroxyapatite (nano-HAP)-containing toothpastes and cream to relieve dentin hypersensitivity, comparing it with those of a commercial desensitizing dentifrice containing calcium sodium phosphosilicate (Novamin® technology) and a standard fluoride dentifrice containing 1,500 ppm fluoride as sodium monofluorophosphate (MFP).

DETAILED DESCRIPTION:
This is a double-blind, randomized, controlled, parallel group, outpatient clinical trial, involving a total of 270 patients diagnosed with dentin hypersensitivity, who will be randomly assigned to nine treatment groups of 30 patients each. Males or females of age 18 to 80 years will be enrolled. The nine groups will be randomly assigned to use one of the nine test products: (1) toothpaste containing nano-HAP (high concentration); (2) toothpaste containing nano-HAP (low concentration); (3) toothpaste containing nano-HAP and potassium nitrate (KNO3); (4) toothpaste containing NovaMin; (5) standard fluoride toothpaste with 1500 ppm MFP; (6) toothpaste containing nano-HAP (medium concentration); (7) placebo toothpaste; (8) cream containing nano-HAP; (9) placebo cream. Subjects will be instructed to use the study toothpaste as their sole oral hygiene product for the 8 weeks treatment duration while the cream will be applied with a retainer tray for 5 minutes before bed at night. For those using toothpastes, subjects will be instructed to brush their teeth twice daily for 2 minutes, morning and last thing before bed, applying on each occasion a one-inch strip of their assigned toothpaste on a wetted commercially available soft-bristled toothbrush. Dentin hypersensitivity examination, which will include air blast sensitivity and cold thermal sensitivity combined with visual analog scale and Dental Pain Scale, will be conducted at baseline, 2, 4, 6, and 8 weeks. Subjects will be screened for adverse effects on every visit, and all observed adverse events will be recorded when they occur.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18 and 80, inclusive
* Must be in good general health based on medical history and oral soft and hard tissue examinations
* Must be willing and able to provide informed consent
* Must be able to read and comprehend study materials
* Must have access to a phone for regular study contact
* Must be willing to use the assigned products according to instructions, and be availability for appointments.
* Must have been diagnosed of having dentin hypersensitivity by a dentist, with at least one sensitive tooth with demonstrated cervical erosion/abrasion or gingival recession
* As a final entrance criteria, the sensitive tooth must respond to:

  * air sensitivity, with Schiff score >1, assessed by use of a one-second blast of air.
  * thermal sensitivity, assessed with frozen cotton pellet, with a pain rating of at least moderate pain on the Dental Pain Scale (DPS) and a score between 30 and 80 mm on a 100 mm scale on the Visual Analog Scale (VAS).

Exclusion Criteria:

* Subjects who answer YES to any of the following questions will not be enrolled into the study:

  * Any history of significant adverse effects following use of oral hygiene products such as toothpastes and mouthwashes?
  * Does the subject have any physical limitations or restrictions that might preclude use of normal oral hygiene procedures (i.e., toothbrushing, mouthrinsing, etc.)?
  * The sensitive tooth is associated with concomitant oral pain due to any other condition such as: soft-tissue lesions or toothache from other dental conditions like dental caries, etc?
  * Has the subject ever reported allergy to drugs or chemicals used in the trial?
  * The sensitive tooth is associated with a periodontal abscess as diagnosed from an X-ray or clinical examination of the tooth?
  * Will the subject receive dental treatment which may affect their participation (i.e. oral prophylaxis)?
  * The sensitive tooth is associated with mobility > 1?
  * Did the subject participate in a dental clinical trial involving oral care products within the past 30 days?
  * Is the subject pregnant, nursing or planning to become pregnant during the course of the study (self-reported)?
  * Does the subject have other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with trial participation or may interfere with the interpretation of trial result and, in the judgment of the investigator, would make the subject inappropriate for entry into this trial?
  * Does the subject have significant oral soft tissue pathology, based on the dentist's visual examination and at the discretion of the investigator?
  * The sensitive tooth is associated with gum pain from gingivitis, occlusal trauma, thermal or chemical burns?
  * Patients having pain from periodontal related causes but not dentin hypersensitivity?
  * Previous professional desensitizing treatment?
  * Subject use of over-the-counter desensitizing products within the previous 3 months?
  * Subjects using medication which could interfere with the perception of pain?
  * Eating disorders or conditions associated with vomiting?
  * Systemic conditions that are etiologic or predisposing to dentinal hypersensitivity?
  * Excessive dietary or environmental exposure to acids?
  * The sensitive tooth was restored in the preceding 3 months?
  * The sensitive tooth is an abutment tooth for fixed or removable prostheses?
  * The sensitive tooth has extensive restorations or restoration extending into the test area?
  * Patients below 18 years or above 80 years of age?

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bennett T Amaechi, BDS, MS, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- School of Dentistry, University of Texas Health Science Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark GE, Troullos ES. Designing hypersensitivity clinical studies. Dent Clin North Am. 1990 Jul;34(3):531-44. PMID 2197126
- [Background] Gillam DG, Bulman JS, Jackson RJ, Newman HN. Efficacy of a potassium nitrate mouthwash in alleviating cervical dentine sensitivity (CDS). J Clin Periodontol. 1996 Nov;23(11):993-7. doi: 10.1111/j.1600-051x.1996.tb00526.x. PMID 8951626
- [Background] Kakar A. A novel computer program for visual analogue scale (VAS). Journal of Dental Research 88 (Special Issue A): 1952, 2009.
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Orro M, Truong T, De Vizio W, Miller S, Chu TC, Boylan D. Thermodontic stimulator--a new technology for assessment of thermal dentinal hypersensitivity. J Clin Dent. 1994;5 Spec No:83-6. PMID 8534379
- [Background] Schiff T, Dotson M, Cohen S, De Vizio W, McCool J, Volpe A. Efficacy of a dentifrice containing potassium nitrate, soluble pyrophosphate, PVM/MA copolymer, and sodium fluoride on dentinal hypersensitivity: a twelve-week clinical study. J Clin Dent. 1994;5 Spec No:87-92. PMID 8534380
- [Background] Ayad F, Ayad N, Delgado E, Zhang YP, DeVizio W, Cummins D, Mateo LR. Comparing the efficacy in providing instant relief of dentin hypersensitivity of a new toothpaste containing 8.0% arginine, calcium carbonate, and 1450 ppm fluoride to a benchmark desensitizing toothpaste containing 2% potassium ion and 1450 ppm fluoride, and to a control toothpaste with 1450 ppm fluoride: a three-day clinical study in Mississauga, Canada. J Clin Dent. 2009;20(4):115-22. PMID 19831164

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Toothpaste Containing Novamin® Technology: Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Control toothpaste containing Novamin® technology
- Control Toothpaste Containing 1500 Ppm Fluoride as MFP: Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Control toothpaste containing 1500 ppm fluoride as MFP
- Test Toothpaste With Nano-HAP (High Concentration): Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Test toothpaste with nano-HAP (high concentration)
- Test Toothpaste With Nano-HAP (Low Concentration): Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Test toothpaste with nano-HAP (low concentration)
- Test Toothpaste With Nano-HAP and Potassium Nitrate (KNO3): Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Test toothpaste with nano-HAP and KNO3
- Control Toothpaste Without Nano-HAP: Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Control toothpaste without nano-HAP
- Test Toothpaste With Nano-HAP (Medium Concentration): Participants will be instructed to apply a full ribbon of toothpaste to a damp toothbrush. Participants will then brush for 2 minutes followed by rinsing with 15 mL of water. Participants will be instructed not to eat or drink for 30 minutes following brushing. Brushing will be performed twice a day (morning and evening).
  Test toothpaste with nano-HAP (medium concentration)
- Test Cream With Nano-HAP (Higher Concentration): Participants will be instructed to brush for 2 minutes morning and evening with a full ribbon of standard fluoride toothpaste. After the evening brushing, participants will then insert custom-made trays loaded with a full ribbon of cream. Participants will be instructed to remove the trays after 5 minutes and expectorate the cream. Participants will be instructed not to eat or drink until the next morning following cream use.
  Test cream with nano-HAP (higher concentration)
- Control Cream Without Nano-HAP: Participants will be instructed to brush for 2 minutes morning and evening with a full ribbon of standard fluoride toothpaste. After the evening brushing, participants will then insert custom-made trays loaded with a full ribbon of cream. Participants will be instructed to remove the trays after 5 minutes and expectorate the cream. Participants will be instructed not to eat or drink until the next morning following cream use.
  Control cream without nano-HAP
Period: Overall Study
Arm/Group | Control Toothpaste Containing Novamin® Technology | Control Toothpaste Containing 1500 Ppm Fluoride as MFP | Test Toothpaste With Nano-HAP (High Concentration) | Test Toothpaste With Nano-HAP (Low Concentration) | Test Toothpaste With Nano-HAP and Potassium Nitrate (KNO3) | Control Toothpaste Without Nano-HAP | Test Toothpaste With Nano-HAP (Medium Concentration) | Test Cream With Nano-HAP (Higher Concentration) | Control Cream Without Nano-HAP
Started | 21 | 20 | 22 | 22 | 24 | 20 | 22 | 26 | 26
Completed | 20 | 20 | 19 | 22 | 24 | 20 | 22 | 25 | 26
Not Completed | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Toothpaste Containing Novamin® Technology | Control Toothpaste Containing 1500 Ppm Fluoride as MFP | Test Toothpaste With Nano-HAP (High Concentration) | Test Toothpaste With Nano-HAP (Low Concentration) | Test Toothpaste With Nano-HAP and Potassium Nitrate (KNO3) | Control Toothpaste Without Nano-HAP | Test Toothpaste With Nano-HAP (Medium Concentration) | Test Cream With Nano-HAP (Higher Concentration) | Control Cream Without Nano-HAP | Total
Number analyzed (Participants) | 20 | 20 | 19 | 22 | 24 | 20 | 22 | 25 | 26 | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.3 (10.5) | 45.85 (15.76) | 53.6 (11.0) | 52.8 (11.2) | 43.7 (12.8) | 45.35 (11.37) | 47.14 (14.54) | 41.4 (14.14) | 49.38 (10.62) | 47.61 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 18 | 16 | 18 | 13 | 17 | 19 | 22 | 152
  Male | 5 | 6 | 1 | 6 | 6 | 7 | 5 | 6 | 4 | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race Ethnicity: Asian or Pacific Islander | 3 | 0 | 0 | 1 | 0 | 2 | 4 | 1 | 3 | 14
  Race Ethnicity: Black not Hispanic | 1 | 0 | 1 | 2 | 0 | 2 | 1 | 4 | 4 | 15
  Race Ethnicity: Hispanic | 8 | 15 | 13 | 12 | 15 | 10 | 11 | 13 | 14 | 111
  Race Ethnicity: Other | 2 | 0 | 1 | 3 | 2 | 1 | 0 | 0 | 1 | 10
  Race Ethnicity: White not Hispanic | 6 | 5 | 4 | 4 | 7 | 5 | 6 | 7 | 4 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in VAS (Visual Analog Scale) With Air Stimulation
Description: Patient's response to an air stimulus is recorded on a Visual Analog Scale of 0-100 with 0 representing no pain and 100 representing the worst possible pain.
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | Control Toothpaste Containing Novamin® Technology | Control Toothpaste Containing 1500 Ppm Fluoride as MFP | Test Toothpaste With Nano-HAP (High Concentration) | Test Toothpaste With Nano-HAP (Low Concentration) | Test Toothpaste With Nano-HAP and Potassium Nitrate (KNO3) | Control Toothpaste Without Nano-HAP | Test Toothpaste With Nano-HAP (Medium Concentration) | Test Cream With Nano-HAP (Higher Concentration) | Control Cream Without Nano-HAP
Number analyzed (Participants) | 20 | 20 | 19 | 22 | 24 | 20 | 22 | 25 | 26
percentage change from baseline | -51.44 (5.31) | -51.59 (5.57) | -41.59 (8.08) | -38.64 (5.85) | -53.16 (5.99) | -47.19 (7.13) | -56.85 (7.98) | -38.99 (5.37) | -50.67 (4.93)

2. Primary Outcome: Percentage Change From Baseline in VAS (Visual Analog Scale) With Cold Stimulation
Description: Patient's response to cold stimulus is recorded on a Visual Analog Scale of 0-100 with 0 signifying no pain and 100 signifying the worst possible pain
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | Control Toothpaste Containing Novamin® Technology | Control Toothpaste Containing 1500 Ppm Fluoride as MFP | Test Toothpaste With Nano-HAP (High Concentration) | Test Toothpaste With Nano-HAP (Low Concentration) | Test Toothpaste With Nano-HAP and Potassium Nitrate (KNO3) | Control Toothpaste Without Nano-HAP | Test Toothpaste With Nano-HAP (Medium Concentration) | Test Cream With Nano-HAP (Higher Concentration) | Control Cream Without Nano-HAP
Number analyzed (Participants) | 20 | 20 | 19 | 22 | 24 | 20 | 22 | 25 | 26
percentage change from baseline | -48.14 (4.63) | -34.96 (6.97) | -44.71 (4.78) | -31.95 (6.88) | -42.49 (6.70) | -35.67 (5.16) | -48.80 (6.21) | -34.90 (3.4) | -39.36 (4.66)

3. Primary Outcome: Percentage Change From Baseline in DPS (Dental Pain Scale) With Air Stimulation
Description: Patient's response to an air stimulus is recorded on a Dental Pain Scale (none[1]-mild[2]-moderate[3]-severe[4]).
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | Control Toothpaste Containing Novamin® Technology | Control Toothpaste Containing 1500 Ppm Fluoride as MFP | Test Toothpaste With Nano-HAP (High Concentration) | Test Toothpaste With Nano-HAP (Low Concentration) | Test Toothpaste With Nano-HAP and Potassium Nitrate (KNO3) | Control Toothpaste Without Nano-HAP | Test Toothpaste With Nano-HAP (Medium Concentration) | Test Cream With Nano-HAP (Higher Concentration) | Control Cream Without Nano-HAP
Number analyzed (Participants) | 20 | 20 | 19 | 22 | 24 | 20 | 22 | 25 | 26
percentage change from baseline | -35.14 (3.53) | -43.35 (4.39) | -34.15 (4.65) | -38.63 (3.70) | -43.95 (3.62) | -33.63 (4.74) | -49.35 (5.66) | -17.47 (3.22) | -28.54 (3.73)

4. Primary Outcome: Percentage Change From Baseline in DPS (Dental Pain Scale) With Cold Stimulation
Description: Patient's response to an cold stimulus is recorded on a Dental Pain Scale (none[1]-mild[2]-moderate[3]-severe[4]).
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | Control Toothpaste Containing Novamin® Technology | Control Toothpaste Containing 1500 Ppm Fluoride as MFP | Test Toothpaste With Nano-HAP (High Concentration) | Test Toothpaste With Nano-HAP (Low Concentration) | Test Toothpaste With Nano-HAP and Potassium Nitrate (KNO3) | Control Toothpaste Without Nano-HAP | Test Toothpaste With Nano-HAP (Medium Concentration) | Test Cream With Nano-HAP (Higher Concentration) | Control Cream Without Nano-HAP
Number analyzed (Participants) | 20 | 20 | 19 | 22 | 24 | 20 | 22 | 25 | 26
percentage change from baseline | -35.37 (3.54) | -30.18 (4.15) | -39.81 (3.60) | -38.41 (3.88) | -35.03 (3.65) | -34.07 (3.70) | -46.21 (4.22) | -15.30 (2.57) | -25.57 (2.97)

ADVERSE EVENTS:
Time Frame: Baseline to 8 weeks
Arm/Group | Control Toothpaste Containing Novamin® Technology | Control Toothpaste Containing 1500 Ppm Fluoride as MFP | Test Toothpaste With Nano-HAP (High Concentration) | Test Toothpaste With Nano-HAP (Low Concentration) | Test Toothpaste With Nano-HAP and Potassium Nitrate (KNO3) | Control Toothpaste Without Nano-HAP | Test Toothpaste With Nano-HAP (Medium Concentration) | Test Cream With Nano-HAP (Higher Concentration) | Control Cream Without Nano-HAP
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20 | 0/22 | 0/20 | 0/21 | 0/20 | 0/22 | 0/25 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/22 | 0/20 | 0/21 | 0/20 | 0/22 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20 | 0/22 | 0/20 | 0/21 | 0/20 | 0/22 | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No